CLINICAL TRIAL: NCT03147118
Title: Evaluating Palpation Guided Injections in Trapeziometacarpal Arthritis
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00059888
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Injection Site; Arthritis;Hand/Finger(S)
Keywords: trapeziometacarpal arthritis
MeSH Terms: interventions — Arthrography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Arthrogram — Contrast dye will be included in the standard injection of lidocaine and corticosteroid. After injection, the participant will have 2 radiograph views of the thumb.

SUMMARY:
The objective of this study is to evaluate the accuracy of trapeziometacarpal injections using palpation alone. The importance of this study is one of education, cost containment, and decreased risk to the patient. If it can be shown that the accuracy of trapeziometacarpal injections using palpation alone is similar to the reported accuracy of ultrasound and fluoroscopy, then these guided techniques may not be needed.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the accuracy of trapeziometacarpal injections using palpation alone. If it can be shown that the accuracy of trapeziometacarpal injections using palpation alone is similar to the reported accuracy of ultrasound and fluoroscopy, then fluoroscopy and ultrasound guided techniques may not be needed. Due to the expenses associated with medications and testing, it is important to not accrue unnecessary costs if there is no perceived benefit. The investigators plan to enroll 50 patients presenting with trapeziometacarpal joint arthritis who agree to participate. These participants will undergo an injection technique consisting of palpating the base of the thumb and placing the needle into the trapeziometacarpal joint without the guidance of ultrasound or fluoroscopy. Contrast dye will be included in the standard injection of lidocaine and corticosteroid. After injection, the participant will have 2 fluoroscopy views of the thumb. The images will not be evaluated for injection accuracy prior to the patient leaving the clinic, so as to not introduce any bias by the treating physician. These images will be blindly reviewed by three investigators at a later date, and determined by consensus if there is contrast material in the joint. The accuracy rate can then be compared to data regarding accuracy of fluoroscopic and ultrasound guided injections of the trapeziometacarpal joint. If there is a similar accuracy rate between modalities, it can be concluded that ultrasound may not be worth the added cost to the patient and fluoroscopy may not be worth the added cost or radiation to the participant. Additionally, participants will be contacted at 6 weeks post injection to evaluate post-injection arthritis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* The patient has clinical signs of trapeziometacarpal arthritis and are willing to obtain a post injection x-ray
* The patient is over the age of 18 years of age.

Exclusion Criteria:

* The patient has a known allergy to contrast dye
* The patient has a planned surgery on the trapeziometacarpal joint within 6 weeks following injection
* Patients who are pregnant or believe they may be pregnant
* Prisoners
* Patients who are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with trapeziometacarpal arthritis and a treatment plan including intra-articular steroid injections
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of injection | radiograph immediately after injection (<5 mins)
  Accuracy judged in a blinded fashion, rated injection in joint or out of joint

CONTACTS AND LOCATIONS:
Overall Officials: John Sanders, MD, Principal Investigator — Prisma Health-Upstate
Locations (1):
- The Hand Center, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No